CLINICAL TRIAL: NCT04818359
Title: Movement and Health Beyond Care, MoviS: Nutrition and Exercise Educational Programs for Breast Cancer Survivors
Brief Title: Movement and Health Beyond Care (MoviS)
Acronym: MoviS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Urbino "Carlo Bo" (Other)
Collaborators: Presidio Ospedaliero Unico "Santa Maria della Misericordia", Urbino (Unknown); National Cancer Institute, Milan (Other)
Responsible Party: Principal Investigator, Elena Barbieri, Associate Professor, University of Urbino "Carlo Bo"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UniUrb_21/10.07.2019
Record Dates: First submitted 2021-02-22; First posted 2021-03-26 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Survivors
Keywords: Breast Cancer; Exercise; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to undergo either a lifestyle recommendations and supervised exercise program or only lifestyle recommendations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Supervised exercise program: MoviS Training. Lifestyle (nutrition and exercise) counseling based on WCRF 2018 recommendations; psychological well-being counseling which comprises evaluation for anxiety and depression.
  Interventions: Behavioral: MoviS Training
- Control Arm (No Intervention): Lifestyle (nutrition and exercise) counseling based on WCRF 2018 recommendations; psychological well-being counseling which comprises evaluation for anxiety and depression.

INTERVENTIONS:
Behavioral: MoviS Training — Patients will undergo a supervised exercise program consisting of 3 months of aerobic exercise training (2 d/week of directly supervised exercise and 1 d/week of remotely supervised exercise) with a progressive increase in exercise intensity (40-70% of heart rate reserve) and duration (20-60 min).
  Arms: Interventional Arm

SUMMARY:
MoviS is a randomized controlled trial on the effect of aerobic exercise training on quality of life (QoL) among breast cancer (BC) survivors.

Patients randomized to the intervention arm will receive lifestyle recommendations (nutrition and exercise) and will undergo the MoviS Training program, whereas control arm patients will receive lifestyle recommendations. The MoviS Training program consists of 3 months, 3 times per week, aerobic exercise, which will be supervised both directly (2 days each week) and remotely (1 day each week). Exercise intensity (40% to 70% of heart rate reserve) and duration (20 to 60 mins) will be gradually increased throughout the training period. Both arms will receive counseling on psychological well-being.

The primary outcome is the improvement of QoL. The secondary outcome is the improvement of the health-related parameters.

Study variables will be sampled and compared between and within groups at the baseline, after the 3 month intervention period, ad interim in the short term (6 months) and long term (12 and 24 months).

DETAILED DESCRIPTION:
BACKGROUND BC is the most common invasive cancer in women and evidence has shown that exercise can significantly improve the outcomes of BC survivors. MoviS (Movement and Health Beyond Care) is a randomized controlled trial that aims to evaluate the potential health benefits of exercise and proper nutritional habits.

Aim The present research study aims to assess the efficacy of aerobic exercise training on the QoL of high-risk BC survivors and the improvement of health-related factors.

Methods BC patients (sample size n=172), age 30-70 years, non-metastatic, stage 0-III, non-physically active, 6-12 months post-surgery, and post chemo- or radio-therapy, with a high risk of recurrence defined by one or more of the following criteria: BMI ≥ 25, diagnosis of metabolic syndrome, increased level of blood testosterone and insulin will be randomly allocated to the interventional arm (lifestyle recommendations and MoviS Training) or control arm (lifestyle recommendations). The MoviS Training consists of 3 months of aerobic exercise training (2 d/week of directly supervised and 1 d/week of remotely supervised exercise) with a progressive increase in exercise intensity (40-70% of heart rate reserve) and duration (20-60 min). Both arms will receive counseling on healthy lifestyle habits (nutrition and exercise) based on the World Cancer Research Fund (WCRF) 2018 guidelines through the DIANA-Web platform. All patients will also undergo psychological well-being counseling, which comprises evaluation for anxiety and depression.

The primary outcome is the improvement of the QoL assessed by the European Organization for Research and Treatment of Cancer QoL (EORTC QLQ-C30) questionnaire.

The secondary outcome is the improvement of health-related parameters such as: fatigue; anthropometric measurements and body composition; cardiac function indexes and heart rate variability; functional parameters (cardiorespiratory fitness, muscle flexibility and strength, coordination and posture variability, upper limb muscle viscoelastic characteristics); psychological well-being; metabolic, hormonal and inflammatory risk factors; gut microbiota; osteoporosis level; recurrences. Diet habits, physical activity level, pharmacological treatments and comorbidity will be recorded as confounding factors and covariates.

The hypothesis is that supervised exercise may improve QoL and health-related factors of BC survivors with a high risk of recurrence.

Data will be collected at baseline and after the 3 month intervention period, ad interim in the short term (6 months) and long term (12 and 24 months).

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of BC (stage 0-II-III, without metastases or recurrences diagnosis at recruitment).
2. After surgery and chemotherapy and/or radiotherapy treatments.
3. Maximum 12 months from surgical treatment.
4. Minimum 6 months from the end of chemotherapy.
5. Risk of recurrence will be identified with meeting at least 1 of the following criteria: BMI at diagnosis ≥ 25 kg/m2, testosterone ≥ 0.4 ng/mL (for women); serum insulin ≥ 25 µU/mL (170 pmol/L); metabolic syndrome (at least 3 of the following 5 factors): a. glycemia ≥ 100 mg/dL (6.05 mmol/L); b. triglycerides ≥150 mg/dL (1.69 mmol L); c. HDL-C <50 mg/dL (1.29 mmol/L) (woman), <40 mg/dL (1.04 mmol/L) (man); d. waist circumference ≥ 80 cm (woman), ≥ 90 cm (man); e. blood pressure ≥ 130/85 mmHg.
6. Non-physically active: subjects who were not regularly active (assessed by IPAQ) for at least 6 months.

Exclusion criteria:

1. Not suitable for non-competitive physical activity after the cardiological medical examination.
2. Disabling pneumological, cardiological, neurological, orthopedic comorbidities and mental illness that prevent the exercise performance.
3. Treatment with drugs that alter the heart rate response to exercise.
4. Treatment with antidepressant drugs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed by questionnaire | Baseline - after 3, 6, 12, 24 months
  Change in quality of life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Scores ranging from 0 to 100; higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Fatigue | Baseline - after 3, 6, 12, 24 months
  Change in fatigue perception assessed by brief fatigue inventory (BFI) questionnaire. The score of the questionnaire ranges from 0 to 90. A higher score means more severe fatigue.
Anthropometry | Baseline - after 3, 6, 12, 24 months
  Change body mass index (BMI) expressed as body mass (kg) / height2 (m2).
Body composition | Baseline - after 3, 6, 12, 24 months
  Change fat mass (%) assessed by bioelectrical impedance analysis.
Cardiac function indexes | Baseline - after 3, 6, 12, 24 months
  Change in the global longitudinal strain (%) assessed by echocardiography.
Heart rate variability | Baseline - after 3 months
  Change in heart rate variability assessed by 24-Holter monitoring.
Cardiorespiratory fitness | Baseline - after 3, 6, 12, 24 months
  Change in cardiorespiratory fitness assessed by estimated maximal oxygen uptake (mL/min/kg).
Flexibility | Baseline - after 3, 6, 12, 24 months
  Change in muscle flexibility assessed by sit & reach test (m).
Muscular fitness | Baseline - after 3, 6, 12, 24 months
  Change strength assessed by isometric hand grip strength test (kg).
Proprioceptive recalibration | Baseline - after 6 months
  Change assessed by stabilometry (Mean Velocity) (mm2/sec2).
Posture balance | Baseline - after 6 months
  Change assessed by stabilometry (Romberg Quotient test-European variant) (% over or under 100).
Upper limb muscles viscoelastic characteristics | Baseline - after 3 months
  Change in the muscle properties of the pectoralis major, upper trapezius, and sternoclavicular mastoid muscle assessed by a hand-held myotonometer.
Psychological well-being | Baseline - after 3, 6, 12, 24 months
  Change in mood profile assessed by Profile of Mood States (POMS) questionnaire. The POMS questionnaire gives a 5-point Likert scale; a higher score indicates increased negative mood.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) Index | Baseline - after 3, 6, 12, 24 months
  Change in HOMA-IR Index calculated as HOMA-IR = (FPI × FPG)/22.5, where FPI is fasting plasma insulin concentration (mU/l) and FPG is fasting plasma glucose (mmol/L), or as HOMA-IR = (FPI × FPG)/405 if fasting plasma glucose is expressed in mg/dL.
Insulin-like growth factor (IGF-1) | Baseline - after 3, 6, 12, 24 months
  Change in IGF-1 assessed by blood samples (µg/L).
C-reactive protein | Baseline - after 3, 6, 12, 24 months
  Change in high sensitivity C-reactive protein assessed by blood samples (mg/L).
Gut microbiota | Baseline - after 3, 6, 12, 24 months
  Change in microbial diversity (species diversity %) assessed by next-generation sequencing (NGS) of the V3-V4 region of the 16S rDNA gene.
Osteoporosis level | Baseline - after 12 and 24 months
  Change in computerized bone mineralometry assessed by T-Score (Normal: +2.5> T-score> -1.0; Osteopenia: -1.0> T-score> -2.5; Osteoporosis: T-score <-2.5; Severe osteoporosis: T-score <-2.5 with one or more fragility fractures).
Recurrences | Baseline - after 3, 6, 12, 24 months
  Recurrences free interval defined as time from registration to time of documented recurrent disease.

OTHER OUTCOMES:
Diet habits | Baseline - after 3, 6, 12, 24 months
  Change in dietary intake assessed by questionnaire (14-item Mediterranean diet adherence screener, MEDIET) through DIANAWeb platform. Higher levels (8-9, or >10 points in the 14-item score) indicates adherence to the Mediterranean diet.
Physical activity level | Baseline - after 3, 6, 12, 24 months
  Change in physical activity level assessed by the sensewear armband activity monitor and by the international physical activity questionnaire (IPAQ). The output of both assessments expressed in metabolic equivalents (METs)-min/week.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Presidio Ospedaliero Unico "Santa Maria della Misericordia", Urbino, Urbino, PU
  - University of Urbino Carlo Bo, Urbino, PU

REFERENCES:
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107
- [Derived] Donati Zeppa S, Natalucci V, Agostini D, Vallorani L, Amatori S, Sisti D, Rocchi MBL, Pazienza V, Perri F, Villani A, Binda E, Panebianco C, Mencarelli G, Ciuffreda L, Ferri Marini C, Annibalini G, Lucertini F, Bartolacci A, Imperio M, Virgili E, Catalano V, Piccoli G, Stocchi V, Emili R, Barbieri E. Changes in gut microbiota composition after 12 weeks of a home-based lifestyle intervention in breast cancer survivors during the COVID-19 lockdown. Front Oncol. 2023 Sep 1;13:1225645. doi: 10.3389/fonc.2023.1225645. eCollection 2023. PMID 37727203
- [Derived] Natalucci V, Ferri Marini C, De Santi M, Annibalini G, Lucertini F, Vallorani L, Panico AR, Sisti D, Saltarelli R, Donati Zeppa S, Agostini D, Gervasi M, Baldelli G, Grassi E, Nart A, Rossato M, Biancalana V, Piccoli G, Benelli P, Villarini A, Somaini M, Catalano V, Guarino S, Pietrelli A, Monaldi S, Sarti D, Barocci S, Flori M, Rocchi MBL, Brandi G, Stocchi V, Emili R, Barbieri E. Movement and health beyond care, MoviS: study protocol for a randomized clinical trial on nutrition and exercise educational programs for breast cancer survivors. Trials. 2023 Feb 22;24(1):134. doi: 10.1186/s13063-023-07153-y. PMID 36814313